CLINICAL TRIAL: NCT05268237
Title: A Phase Ib/IIa, Single Ascending Dose Study of the Safety, Tolerability and Preliminary Efficacy of Sublingual Liraglutide in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability and Preliminary Efficacy of Sublingual Liraglutide in Patients With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biolingus (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIOL-001
Record Dates: First submitted 2022-02-16; First posted 2022-03-07 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is being conducted in 2 parts. Part 1 is an open-label study with no requirements for randomisation or blinding. Part 2 is a placebo-controlled, observer blinded, partially randomised, repeated treatment double-blinded controlled trial with active comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Open Label (Experimental): Part 1 of the trial will utilise an open label, single ascending dose, repeated treatment design. It will involve 3 subjects, each of whom will receive three single ascending doses of SL liraglutide (3, 12, 30mg and subcutaneous (SC) liraglutide (active comparator) with a mixed meal tolerance test (MMTT), separated by 1 week washout between doses.
  Interventions: Drug: Liraglutide
- Part 2: Investigator blind (Experimental): Part 2 of the trial will utilise an investigator-blind, sponsor open, placebo-controlled, randomised, repeated treatment study design. It will involve 12 subjects. Each subjects will receive one of three possible doses of SL-liraglutide (to be decided by the Safety Monitoring Committee following analysis of the results from Part 1), SL-placebo or SC liraglutide in a randomised order with MMTT separated by 1 week washout between doses.
  Interventions: Drug: Liraglutide; Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Sublingual or subcutaneous liraglutide
Drug: Placebo — Sublingual placebo
  Arms: Part 2: Investigator blind

SUMMARY:
This is a phase Ib/IIa, single ascending dose study of the safety, tolerability and preliminary efficacy of sublingual (SL) Liraglutide in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This Phase Ib/IIa study of SL liraglutide will be conducted at the Phase 1 Clinical Trial Center, Prince of Wales Hospital, Hong Kong. Study subjects will be patients with T2DM who have not previously received liraglutide. The study seeks to document the utility of a SL formulation of the approved active ingredient liraglutide, currently marketed in a subcutaneous (SC) formulation as Victoza®.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-65 years (inclusive)
2. Body mass index (BMI) 18-35 kg/m2, inclusive
3. Normal blood pressure or well managed hypertension (systolic blood pressure <160mmHg, diastolic blood pressure <100 mmHg)
4. Confirmed diagnosis of T2DM (by repeated laboratory findings) for at least 1 year.
5. Subjects under glycemic control on a stable dose of metformin (within the standard of care dose range up to 2 g daily) for at least 2 months prior to enrolment or those who manage their condition only by diet/exercise.
6. For subjects on a stable dose of concomitant metformin for at least 2 months prior to enrolment, the subject's dose of metformin will be required to remain constant until at least the completion of MMTT on the final dosing day. Subjects whose concomitant glucose lowering medication changes during the dosing phase of the study will be discontinued and may be replaced.
7. For subjects not in receipt of concomitant metformin for at least 2 months prior to enrolment, and who manage their condition only by diet/exercise, documentation of stable glycemic control under current condition management for at least 2 months prior to enrolment, as confirmed by HbA1c. For subjects who meet this criterion, no change in disease management is permitted until at least the completion of MMTT on the final dosing day. Any subject who requires a change in disease management, including initiation of any diabetes medication during the study, will be discontinued from the study and may be replaced.
8. Fasting plasma glucose ≥5.6 mmol/L at screening
9. HbA1c ≥6.5% and ≤9.0% at screening
10. Vital signs after 10 minutes resting supine:

    1. 90 mmHg <systolic blood pressure <160 mmHg
    2. 40 mmHg <diastolic blood pressure <100 mmHg
    3. 40 bpm <heart rate <100 bpm Duplicate assessments will be performed and the average of the two assessments of blood pressure will be used.
11. Standard 12-lead ECG parameter results at screening, after 10 minutes resting in supine position, within 120 ms <PR <220 ms, QRS <120 ms, QTcF ≤450 ms (males), QTcF ≤470 ms (females).
12. No history of significant cardiovascular disease over the preceding 3 years or any other major disease other than T2DM and well managed hypertension, unless permitted at the discretion of the PI.
13. Negative test for selected drugs of abuse at screening (does not include alcohol) and at admission (testing at admission does include alcohol breath test). A positive result may be verified by re-testing (up to one false positive result permitted) and may be followed up at the discretion of the PI.
14. Females must be non-pregnant and non-lactating, and either surgically sterile for a minimum of 6 months (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use highly effective contraceptive method (oral contraceptives pills, long-acting implantable hormones, injectable hormones, a vaginal ring or an intrauterine device [IUD]) from screening until study completion, or be post-menopausal for ≥12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels (≥ 40 IU/mL) at screening for amenorrheic female subjects. Females who are abstinent from heterosexual intercourse will also be eligible.
15. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and admission and be willing to have additional pregnancy tests as required throughout the study.
16. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the subject and his partner must be surgically sterile (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from screening until study completion. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner (WOCBP), as per Inclusion Criterion #14. Male subjects whose female partner is post-menopausal, and subjects who are abstinent from heterosexual intercourse will also be eligible. Male subjects must agree to refrain from donating sperm from screening until study completion.

Exclusion Criteria:

1. Pregnant or lactating, or intending to become pregnant within 30 days after last dose of study drug.
2. Participation in a clinical trial within 30 days before enrolment; use of any experimental oral therapy within 30 days or 5 half-lives prior to enrolment, whichever is greater; or use of any biologic therapy within 12 weeks or 5 half-lives prior to enrolment, whichever is greater. Subjects who have received an experimental therapy that has no half-life, such as a vaccine, should have completed that therapy at least 30 days prior to enrolment.
3. Any vaccine 2 weeks prior to first study drug administration until 2 weeks after the last dose, with the exception of current seasonal influenza vaccination.
4. Use of any weight loss agent within the preceding 4 weeks.
5. Surgery or hospitalization during the 4 weeks prior to screening.
6. Planned procedure or surgery during the study.
7. Blood transfusion within 8 weeks prior to screening.
8. Donation or loss of blood (excluding the volume of blood that will be drawn during screening procedures) as follows: ≥ 300 mL of blood within 30 days prior to study drug administration.
9. Poor peripheral venous access.
10. Alcohol and/or substance abuse or dependence within the past 2 years.
11. Within the last 2 years, unstable or clinically significant cardiovascular disease (e.g. myocardial infarction, angina pectoris, New York Heart Association Class II or more cardiac failure).
12. History of pancreatitis
13. History or presence of an abnormal ECG that is clinically significant in the PI's opinion and/or evidence of prior myocardial infarction within 2 years before screening.
14. History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease, coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g. hypokalemia, hypomagnesemia, hypocalcaemia), or family history of sudden unexplained death or long QT syndrome.
15. Impaired hepatic function as indicated by screening aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 x or total bilirubin ≥ 1.5 x the upper limit of normal (ULN), which remains above these limits if retested due to a slightly elevated initial result or abnormalities in synthetic function tests that are judged by the PI to be clinically significant.
16. Unstable hypo- or hyperthyroidism.
17. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome Type 2.
18. Current or history of bulimia or anorexia nervosa.
19. History of severe allergy (requiring hospital care), severe reaction to any drug, or any known or suspected allergies or sensitivities to the study drug constituents.
20. Diagnosis with Type 1 Diabetes Mellitus (T1DM) or any previous episodes of diabetic ketoacidosis.
21. History of or ongoing inflammatory bowel disease or diabetic gastroparesis.
22. Severe hypoglycaemia resulting in seizure/unconsciousness/coma/hospitalization in the last 3 months before screening.
23. Persistent hyperglycaemia not controlled by metformin/diet/exercise.
24. Proliferative retinopathy, nephropathy or renal impairment (<60 mL/min as calculated by the CKD-EPI equation) if deemed clinically significant by the PI.
25. Any other serious medical condition, or abnormality in clinical laboratory tests, that would preclude the subject's safe participation in and completion of the study or increase the expected risk of exposure to the investigational product (IP) or would be expected to interfere with the planned evaluations, in the judgment of the PI.
26. Use of diabetes medication other than metformin at screening and between screening and Day 1 assessments.
27. Any medication during the treatment period and within 14 days before first dosing unless permitted by the inclusion criteria or permitted at the discretion of the PI and when the intake is unlikely to interfere with insulin/glucose control.
28. Use of dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 [GLP-1] agonists, sodium glucose transporter 2 inhibitors, insulin, thiazolenindiones, acarbose in the 3 months prior to study enrolment will not be permitted.
29. Unwilling or unable to follow protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events | Through study completion, an average of 6 weeks
  The primary objective of the study is to evaluate the safety and tolerability of single ascending doses of SL liraglutide in subjects with Type II Diabetes Mellitus (T2DM), and the primary outcome measures are therefore the incidence, nature and severity of adverse events, including those that are serious, dose limiting or of special interest.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) for glucose | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Area under the plasma concentration versus time curve (AUC) for glucose | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Peak Plasma Concentration (Cmax) for C-peptide | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Peak Plasma Concentration (Cmax) for insulin | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Area under the plasma concentration versus time curve (AUC) for C-peptide | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Area under the plasma concentration versus time curve (AUC) for insulin | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Insulin secretion rate (ISR) | 5 hours following administration of the study drug
  A secondary objective is to document the pharmacodynamic effect of SL liraglutide through a mixed meal tolerance test (MMTT) following single ascending dosing in treated subjects.
Serum concentration of liraglutide | 5 hours following administration of the study drug
  A secondary objective is to determine the pharmacokinetics (PK) of SL-liraglutide in plasma following single ascending dosing in treated subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine YK Chow, Principal Investigator — Chinese University of Hong Kong; Juliana CN Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Clinical Trials Unit, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.